CLINICAL TRIAL: NCT06027346
Title: A Phase I Study of BIO-008 Injection for Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity in Patients With Advanced Solid Tumors
Brief Title: A Study of Bio-008 in Subjects With Advanced or Metastatic Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BIO-008ONC1001
Record Dates: First submitted 2023-08-14; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor, Adult
Keywords: Tolerance; Pharmacokinetic characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Bio-008 0.3mg/kg (Experimental): group1
  Interventions: Biological: Bio-008
- Bio-008 1.0mg/kg (Experimental): group2
  Interventions: Biological: Bio-008
- Bio-008 3.3mg/kg (Experimental): group3
  Interventions: Biological: Bio-008
- Bio-008 10.0mg/kg (Experimental): group4
  Interventions: Biological: Bio-008
- Bio-008 20.0mg/kg (Experimental): group5
  Interventions: Biological: Bio-008
- Bio-008 30.0mg/kg (Experimental): group6
  Interventions: Biological: Bio-008
- Bio-008 40.0mg/kg (Experimental): group7
  Interventions: Biological: Bio-008

INTERVENTIONS:
Biological: Bio-008 — The subjects in each dose group received the corresponding dose of BIO-008 monotherapy, administered intravenously (ivd) for a duration of 0.5 to 3 hours (the researchers can adjust the administration time according to the patient's tolerance). If there is an infusion reaction, the infusion can be suspended and completed within 12 hours. Administer on the first day of each cycle, once every 3 weeks (1 cycle, i.e. 21 days) (Q3W) until the criteria for termination of treatment or withdrawal from the study are met, whichever occurs first.

SUMMARY:
Phase 1: Dose escalation study (Phase Ia)

Main purpose:

Evaluate the safety and tolerability of BIO-008 in patients with advanced solid tumors, and determine the maximum tolerable dose (MTD) and dose limiting toxicity (DLT) of BIO-008.

Secondary purpose:

Evaluate the pharmacokinetic (PK) characteristics of BIO-008;

Evaluate the immunogenicity of BIO-008.

Exploratory purposes:

Preliminary evaluation of the anti-tumor activity of BIO-008 (if available);

Detect the expression of CLDN18.2 in tumor tissue and explore its correlation with BIO-008 anti-tumor activity indicators (only applicable to subjects who can provide fresh or archived tumor tissue samples before the first administration).

Phase 2: Dose Extension Study (Phase Ib)

Main purpose:

• Preliminary evaluation of ORR of BIO-008 in patients with CLDN18.2 positive advanced gastric cancer or gastroesophageal junction cancer (GC/GEJ), pancreatic cancer (PC) and other solid tumors;

Determine the recommended dose for clinical phase II (RP2D).

Secondary purpose:

Evaluate the safety and tolerability of BIO-008;

Evaluate the PK characteristics of BIO-008;

Evaluate the immunogenicity of BIO-008;

• Evaluate other anti-tumor activity indicators of BIO-008 in patients with CLDN18.2 positive advanced gastric cancer or gastroesophageal junction cancer, pancreatic cancer and other solid tumors;

Evaluate the correlation between the anti-tumor activity of BIO-008 and the expression of CLDN18.2.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed informed consent (ICF) and follow protocol requirements
2. Age is 18~75 years old (including the boundary value), gender is not limited
3. Patients with advanced solid tumors who have histologically or cytologically confirmed standard therapy failure (progressive treatment or intolerance), or no standard therapy regimen, or who are not suitable for standard therapy at this stage
4. Dose escalation study (Phase Ia): Participants agreed to provide fresh or archived tumor tissue samples for assessment of CLDN18.2 expression levels before the first dose (central laboratory), and subjects enrolled in Phase Ia did not require positive CLDN18.2 expression. If the subject cannot provide samples or a sufficient number of slices, he may be evaluated by the investigator if other entry criteria are met
5. Dose extension study (Phase Ib): The subject agreed to provide fresh or archived tumor tissue samples for the assessment of CLDN18.2 expression levels (before the central laboratory) and tested positive for CLDN18.2 by the central laboratory
6. According to RECIST v1.1 standard, dose escalation studies (Phase Ia) have at least evaluable lesions; Dose extension study (Phase Ib) with at least one measurable lesion;
7. The ECOG physical strength score is 0-1 point
8. The estimated survival time is not less than 3 months
9. The toxicity of previous anti-tumor therapy has recovered to grade 1 as defined by CTCAE v5.0 (except for asymptomatic laboratory abnormalities, such as elevated ALP test, hyperuricemia, elevated blood glucose, etc.

   except for toxicity without safety risk judged by the investigator, such as hair loss, pigmentation, grade 2 peripheral neurotoxicity, thyrotoxicity after immune checkpoint inhibitor treatment, except for those who have been controlled after hormone replacement therapy)
10. Within 7 days before the first dose, the functional levels of the bone marrow reserve and organs must meet the following requirements: Bone marrow reserve: Absolute neutrophil count (ANC) 1.5 109 / L, platelet count (PLT) 90109 / L, hemoglobin (HGB)> 90 g / L (no blood transfusion or hematopoietic stimulating factor therapy within 14 days) Coagulation function: activated partial prothrombin time (APTT) extended 1.5 upper limit of normal (ULN), international standardized ratio (INR) 1.5 Liver function: total bilirubin 1.5 ULN (direct bilirubin normal Gilbert syndrome can be enrolled), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 2.5 ULN (if liver metastases, ALT and AST 5 ULN) Renal function: creatinine clearance of 60 mL/min (using the Cockcroft-Gault formula, see Appendix 1) or serum creatinine of 1.5 ULN Qualified fertile patients (men and women) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence, etc.) with their partner during the trial and at least 6 months after the last dose
11. Qualified patients (male and female) with fertility must agree to use reliable contraceptive methods (such as hormone or barrier methods or abstinence) with their partners during the trial period and at least 6 months after the last medication; Female patients of childbearing age must have a negative serum pregnancy test within 7 days before the first use of the investigational drug.

Exclusion Criteria:

1. Allergic or hypersensitivity to similar products or excipients
2. Received other clinical trial drug or treatment within 28 days prior to the first dose
3. They had received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy and immunotherapy within 28 days before the first dose. Enrollment may be judged by the investigator if:

1) Small local palliative radiotherapy (bone metastasis radiotherapy for pain control), more than 14 days since the first dose 2)Use of oral drugs, including fluorouracil and small molecule targeted drugs, more than 14 days or more than 5 half-lives since the first drug administration (whichever is longer) 3) It has been more than 14 days since the first administration of traditional Chinese medicine with anti-tumor indications 4) Nitrosourea or mitomycin C was used more than 6 weeks from the first administration.

4: Have received antitumor drugs for the CLDN18.2 target

5: Vaccination of any live vaccine within 28 days before the first dose (e. g., vaccines against infectious diseases, such as influenza, varicella, or COVID-19, etc.)

6: Those who have received immunosuppressive agents or systemic corticosteroids (receiving more than 10mg of prednisone or equivalent glucocorticoids per day) within 14 days prior to the first dose

7: Major organ surgery or interventional therapy (excluding tumor biopsy, puncture, etc.) or significant trauma within 28 days before the first dose, or required elective surgery during the trial

8: Those who are using anticoagulants, vitamin K antagonists, or heparin treatment may receive prophylactic doses

9: Patients with gastrointestinal obstruction or persistent recurrent vomiting (defined as 3 vomiting at 24 hours) or uncontrolled / severe gastrointestinal bleeding or ulcer within 28 days prior to the first dose

10: Patients with active infection within 1 week prior to the first dose and currently requiring systemic anti-infection treatment

11: Patients with central nervous system metastasis or meningeal metastasis, or other evidence that CNS metastasis or meningeal metastasis has not been controlled and are not eligible by the investigator

12: Poor controlled pleural effusion, pericardial effusion or ascites requiring repeated drainage were judged by the investigator as not suitable for enrollment

13: Patients with a history of interstitial pneumonia, pulmonary fibrosis, radiation pneumonia or interstitial lung disease / pneumonia caused by drugs, as judged by the investigator

14: History of severe cardiovascular and cerebrovascular diseases, including but not limited to:

1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, -degree atrioventricular block, etc.
2. QT interval extension (Fridericia corrected QT value (QTc)> 450 msec in men or> 470 msec in women)
3. Left ventricular ejection fraction was <50%
4. Thromboembolic events requiring therapeutic anticoagulation, or subjects with venous filters
5. According to the New York Cardiology Association (NYHA) standard, grade III to IV cardiac dysfunction
6. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other serious cardiovascular and cerebrovascular events within 6 months prior to the first dose
7. Clinically uncontrolled hypertension (systolic blood pressure 150 mmHg and / or diastolic blood pressure 100mmHg after drug treatment)
8. Any factor that increases the risk of QTc prolongation or arrhythmia, such as hypokalemia with poorly controlled hypokalemia, congenital long QT syndrome, use of any concomitant medication known or potentially prolonged QT interval (see Appendix 4)

15: Patients with a second primary tumor within 5 years before the first dose, except for the following conditions: radical treatment of skin basal cell carcinoma, squamous epithelial cell carcinoma of the skin, or radical resection of carcinoma in situ

16: Previous history of immunodeficiency, including other acquired or congenital immunodeficiency diseases, or a history of organ transplantation, or a history of allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation, or active autoimmune diseases and inflammatory diseases

17: HIV Infection, active HBV infection (HBV DNA 2000 IU / mL or 1104 copies / mL), active HCV infection (HCV RNA above the upper limit of normal), active syphilis infection (positive for syphilis-specific antibody)

18: A known history of substance abuse

19: People with mental illness disorders or poor compliance

20: Unable to tolerate venous blood collection

21: Female patients during pregnancy or lactation

22: The subject was not eligible for the clinical study in the opinion of a history of other serious systemic disease or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE)/severe adverse events (SAE) | from the start of the medication to the end of the study or 28 days after cessation of medication
  To evaluate the safety of Bio-008
Incidence of dose limiting toxicity (DLT) | From day 1 to day 21 after the first dose
  To collect dose limiting toxicities (DLTs) occurring within 21 days after the first dose
Maximum Tolerated Dose (MTD） | From day 1 to day 21 after the first dose
  The maximum tolerated dose (MTD) is commonly estimated to be the maximum dose that can be determined through DLT of two among 6 subjects administered with Bio-008 once every 3 weeks in 21 days cycles.
Objective response rate (ORR) (RECIST 1.1) | From date of randomization until the date of first documented progression, up to 3 months
  These measure are defined as the proportion of subjects with complete response (CR) or partial response (PR)
Recommended Phase 2 Dose (RP2D) | From day 1 to day 21 after the first dose
  The RP2D will be determined during the dose expansion stage of the study. RP2D will be determined using available safety and efficacy data.

SECONDARY OUTCOMES:
Area under plasma concentration vs time curve (AUC) | from the start of the medication to the end of the study or 28 days after cessation of medication
  Changes in AUC over time in participants
Peak plasma concentration (Cmax) | from the start of the medication to the end of the study or 28 days after cessation of medication
  Cmax is the maximum plasma concentration
Time to maximum observed plasma concentration(Tmax) | from the start of the medication to the end of the study or 28 days after cessation of medication
  Tmax is the time in hrs/days it takes to reach Cmax after dosing
Terminal elimination half life (T1/2) | from the start of the medication to the end of the study or 28 days after cessation of medication
  Time for the plasma level of Bio-008 to decrease b y 1/2 during the terminal elimination phase
Immunogenicity | from the start of the medication to the end of the study or 28 days after cessation of medication
  by measurement of Incidence of anti-drug antibodies (ADA) and neutralizing antibody（Nad）
Disease control rate (DCR) (RECIST 1.1) | From date of randomization until the date of first documented progression, up to 3 months
  These measure are defined as the proportion of subjects with CR, PR and stable disease (SD)
Duration of response (DOR) (RECIST 1.1) | From date of randomization until the date of first documented progression, up to 3 months
  These measure are defined as the duration from the first occurrence of confirmed CR or PR until the date of disease progression or death (from any cause)
Progression free survival (PFS) (RECIST 1.1) | From date of randomization until the date of first documented progression, up to 3 months
  These measure are defined as time from start of treatment to tumor progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: gang Ji, PI, Principal Investigator — The First Affiliated Hospital of the Chinese People's Liberation Army Air Force Military Medical University
Locations (1):
- The First Affiliated Hospital of the Chinese People's Liberation Army Air Force Military Medical University, Xi'an, Shaanxi, China